CLINICAL TRIAL: NCT03634566
Title: Effect of N_Acetylcysteine on Liver Functions in Donors in Living Donor Liver Transplantation
Brief Title: Effect of N_Acetylcysteine on Liver Functions in Donors in Living Liver Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Lecturer of anesthesia,intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R 10/2018
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-10

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC group (Active Comparator): Group NC received NAC 150 mg/kg diluted in 100 ml glucose 5 % over 40 minutes followed by NAC 12.5 mg/kg in 500 ml glucose 5% over 4 hours, followed by NAC 6.25 mg/kg for 2 postoperative days
  Interventions: Drug: N-Acetylecysteine
- Control group (Placebo Comparator): Group C (Control group) will receive ringer acetate continuous infusion at same rate for 2 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylecysteine — N-Acetylecysteine 150 mg/kg diluted in 100 ml glucose 5 % over 40 minutes followed by NAC 12.5 mg/kg in 500 ml glucose 5% over 4 hours, followed by NAC 6.25 mg/kg for 2 postoperative days
  Arms: NAC group
Drug: Placebo — Ringer acetate continuous infusion at the same rate for 2 days.
  Arms: Control group

SUMMARY:
our practice for the past 10 years we have noticed a transitional impairment of liver function (elevated liver enzymes, total and direct bilirubin, and elevated serum lactate levels) following donors' liver resection. Several drugs have been investigation on liver regeneration , proven benefit of N-Acetylcysteine (NAC) on rats with steatohpatitis

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II donors
* healthy adult

Exclusion Criteria:

* kidney, liver disease
* any contraindications for organ donation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Serum lactate | 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided